CLINICAL TRIAL: NCT05855928
Title: Effectiveness of Electrical Stimulation and Mime Therapy Versus Electrical Stimulation and PNF Technique Among Bells Palsy Patients
Brief Title: Effectiveness of ES and MT VS ES and PNF Technique Among Bells Palsy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/526
Record Dates: First submitted 2023-03-18; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Bell Palsy
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical Stimulation and Mime Therapy (Other)
  Interventions: Diagnostic Test: Mime Therapy
- Electrical Stimulation and PNF Technique (Experimental)
  Interventions: Diagnostic Test: PNF Technique

INTERVENTIONS:
Diagnostic Test: Mime Therapy — electrical stimulation with the MIME therapy and protocol
  Arms: Electrical Stimulation and Mime Therapy
Diagnostic Test: PNF Technique — electrical stimulation with the PNF technique with the routine physical therapy
  Arms: Electrical Stimulation and PNF Technique

SUMMARY:
To determine the effectiveness of electrical stimulation with MIME therapy versus electrical stimulation with PNF technique for improving strength & restoring lost motor function in the patients of Bell's palsy

ELIGIBILITY:
Inclusion Criteria:

* • Acute, unilateral, lower motor neuron bells palsy patient with house-backmann scale 4

  * Acute onset 1-3 weeks
  * Age group 20-40 years
  * Who were are willing to be a part of the study
  * Patients with the Bell's palsy (Facial paralysis , idiopathic facial paralysis and the herpetic facial paralysis)

Exclusion Criteria:

* • Patient who had the autoimmune disorder, tumors, recent head injury

  * The subject long with the surgery for ear and the fascial nerve palsy
  * Metal dental implants, and pregnant women
  * The patient with any peripheral vascular diseases
  * Central fascial palsy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Facial disability index(FDI) Scale | 6 Months
  Physical function, Difficulties

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University CRC, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No